CLINICAL TRIAL: NCT05226689
Title: A Prospective, Multicenter, RSA Study of the Porous Tibia Baseplate W/Jrny Lock
Brief Title: Porous Baseplate in Total Knee Replacement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Radiostereometric Analysis Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2021:110
Record Dates: First submitted 2022-01-03; First posted 2022-02-07 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- POROUS TIBIA BASEPLATE W/ JRNY LOCK (Other): Fixed-bearing POROUS TIBIA BASEPLATE W/ JRNY LOCK and a Legion cruciate-retaining High-Flex or Deep-dish XLPE tibial insert.
  Interventions: Device: POROUS TIBIA BASEPLATE W/ JRNY LOCK

INTERVENTIONS:
Device: POROUS TIBIA BASEPLATE W/ JRNY LOCK — Fixed-bearing POROUS TIBIA BASEPLATE W/ JRNY LOCK and a Legion cruciate-retaining High-Flex or Deep-dish XLPE tibial insert

SUMMARY:
This is a multi-centre single cohort trial of patients undergoing cruciate-retaining total knee arthroplasty with the Advance Porous fixed bearing tibial baseplate and compatible femoral, patellar, and bearing components.

DETAILED DESCRIPTION:
All patients will undergo post-operative model-based RSA to identify migration of the tibial baseplate with respect to the bone as well as migration of the patellar and femoral components with respect to the bone during the first 2 post-operative years. Patient health and functional outcomes will be recorded at pre- and post-operative intervals for all patients. Peri-operative adverse events and other clinical complications will be captured as encountered.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the knee indicating primary unilateral total knee arthroplasty
* Sufficient ligamentous function to warrant retention of the posterior cruciate ligament
* Aged 21 years or older
* Patients willing and able to comply with follow-up requirements and self-evaluations
* Ability to give informed consent

Exclusion Criteria:

* Active or prior infection
* Medical condition precluding major surgery
* Known medical condition limiting patient life expectancy to < 2 years
* Expected to receive contralateral TKA within 1 year
* Inflammatory arthropathy
* Prior patellectomy
* PCL deficiency
* Major (>25 degree) coronal plane deformity
* Bilateral coronal plane deformity requiring simultaneous bilateral TKA
* Bone defects requiring augments, cones and/or stemmed implants
* Body Mass Index greater than 40

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change between 6 months and 1-year post-operative - tibial baseplate stability | 6 Months and 1 Year
  Maximum total point motion (MTPM) migration of the POROUS TIBIA BASEPLATE W/ JRNY LOCK between 6 months and 1 year post-operative (mm)

SECONDARY OUTCOMES:
Change between 1- and 2-years post-operative - tibial baseplate stability | 1 Year and 2 Years
  Maximum total point motion (MTPM) migration of the POROUS TIBIA BASEPLATE W/ JRNY LOCK between 1 year and 2 years post-operative (mm)
Total MTPM migration of the baseplate at 1 year | 1 Year
  Assessment of the stability of the tibial baseplate (mm)
Establish the post-operative migration pattern of the patellar and femoral components | 6 Weeks and 6 Months
  Assessment of the migration pattern (mm)
What is the magnitude of baseplate displacement that results from patient weight-bearing (single leg stance) versus non-weight-bearing at 1-year post-operation? | 1 Year
  Assessment of the baseplate displacement differences between standing and supine RSA (mm)
European Quality of Life (EQ-5D-5L) | Preoperative, 6 Weeks, 6 Months, 1 Year and 2 Years
  EQ5D consists of 5 subscales; Mobility, Self-care, Usual activities, Pain/Discomfort and Anxiety / depression. A health state score is obtained based on the responses from 1-5 in each subscale, from which a single index value is calculated representing patients' overall health state. EQ5D includes a so called EQ VAS score which is the patients' self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled "the best health you can imagine" and "the worst health you can imagine".
Patient-reported Outcome: Oxford Knee Score | Preoperative, 6 Weeks, 6 Months, 1 Year and 2 Years
  The Oxford Knee Score (OKS) is a patient self-administered 12-item questionnaire with each question having a Likaert-like response option. Each item is scored from 0 to 4, and the items are summated, with lower total scores indicating poorer performance. The OKS measures pain and general activities of daily living.
Forgotten Joint Score (FJS) | Preoperative, 6 Weeks, 6 Months, 1 Year and 2 Years
  The FJS total score range is 0-100, higher scores indicating the patient is able to forget the joint daily or lower degree of joint awareness.
Knee Injury and Osteoarthritis Outcomes Score (KOOS JR.) | Preoperative, 6 Weeks, 6 Months, 1 Year and 2 Years
  The KOOS JR. was a participant completed questionnaire that consists of 7 questions from 3 subscales: stiffness (1 question), pain (4 questions), and function in daily living (2 questions). Standardized answer options are given (5 Likert boxes) and each question was assigned a score from none (0) to extreme (4).
University of California at Los Angeles (UCLA) Activity Level scale | Preoperative, 6 Weeks, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change in UCLA activity score compared to baseline in the study cohort. UCLA activity scores range from 1 to 10, and is a measure of activity with 10 being most active.
Pain VAS | Preoperative, 6 Weeks, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in patient reported satisfaction as measured using the visual analogue scale (VAS) from 0 (No pain) - 100 (Worst pain imaginable)
Satisfaction VAS | Preoperative, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in patient reported pain severity as measured using the visual analogue scale (VAS) from 0 (Unsatisfied) - 100 (Completely satisfied)
Patient complications | 6 Weeks, 6 Months, 1 Year and 2 Years
  Evaluate the type and frequency of the complications/adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Naudie, MD, Principal Investigator — London Health Sciences Centre
Locations (2):
- Canada (2):
  - Concordia Hospital, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario